CLINICAL TRIAL: NCT05346276
Title: 68Ga-DOTA-hLAG-3 PET Imaging of LAG-3 Expression in Cancers
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital of Xiamen University (Other)
Responsible Party: Sponsor
Other Study IDs: XMYY-2022KY041
Record Dates: First submitted 2022-04-06; First posted 2022-04-26 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2022-12

CONDITIONS: PET/CT; hLAG-3; TUMOR
Keywords: Tumor; PET/CT; diagnosis; hLAG-3
MeSH Terms: conditions — Neoplasms; Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 68Ga-DOTA-hLAG-3 PET/CT: Each participant receives a single intravenous injection of 68Ga-DOTA-hLAG-3, and undergo PET/CT imaging within the specified time
  Interventions: Diagnostic Test: 68Ga-DOTA-hLAG-3 PET/CT

INTERVENTIONS:
Diagnostic Test: 68Ga-DOTA-hLAG-3 PET/CT — Each participant receives a single intravenous injection of 68Ga-DOTA-hLAG-3, and undergo PET/CT imaging within the specified time.

SUMMARY:
To evaluate the potential usefulness of 68Ga-DOTA-hLAG-3 positron emission tomography/computed tomography (PET/CT) for the evaluation of LAG-3 expression in primary and/or metastatic tumors, compared with histopathological results.

DETAILED DESCRIPTION:
Participants with cancer underwent 68Ga-DOTA-hLAG-3 PET/CT for an initial assessment. Tumor uptake was quantified by the maximum standard uptake value (SUVmax) and mean SUV (SUVmean). In addition, the LAG-3 expression of lesions was confirmed by histopathological analyzing. The quantitative parameters of 68Ga-DOTA-hLAG-3 PET/CT were compared with histopathological result to evaluate the diagnostic efficacy.

ELIGIBILITY:
Inclusion Criteria:

* (i) adult patients (aged 18 years or order);
* (ii) patients with newly diagnosed or previously treated malignant tumors (supporting evidence may include magnetic resonance imaging (MRI), CT, tumor markers and pathology report);
* (iii) patients who had scheduled 68Ga-NK224 PET/CT scans;
* (iv) patients who were able to provide informed consent (signed by participant, parent or legal representative) and assent according to the guidelines of the Clinical Research Ethics Committee.

Exclusion Criteria:

* (i) patients with non-malignant lesions;
* (ii) patients with pregnancy;
* (iii) the inability or unwillingness of the research participant, parent or legal representative to provide written informed consent.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients with newly diagnosed or previously treated malignant tumors(supporting evidence may include magnetic resonance imaging (MRI), CT, tumor markers and pathology report)
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2024-12-13 (Actual)

PRIMARY OUTCOMES:
The concordance between 68Ga-DOTA-hLAG-3 PET/CT and histopathological result in LAG-3 expression | 30 days
  For 68Ga-DOTA-hLAG-3 PET/CT parameter, the maximum standard uptake value (SUVmax) is measured by defining a region of interest (ROI) around the primary tumor. For histopathological results, the level of LAG-3 expression is quantified as low (<1%), medium (1-49%), and high (>49%), respectively. Finally, one-way ANOVA tast will be used to test the concordance between 68Ga-DOTA-hLAG-3 PET/CT and histopathological result in LAG-3 expression.

SECONDARY OUTCOMES:
Evaluate the inter-tumor heterogeneity | 30 days
  For the inter-tumor heterogeneity, the investigators will use the Wilcoxon test to compare the SUVmax values of primary tumor and metastases, which are measured by 68Ga-DOTA-hLAG-3 PET/CT, for indirectly evaluating the inter-tumor heterogeneity.

CONTACTS AND LOCATIONS:
Overall Officials: Long Sun, PhD, Study Chair — The First Affiliated Hospital of Xiamen University
Locations (1):
- The First affiliated hospital of xiamen university, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: No